CLINICAL TRIAL: NCT05414513
Title: The Turkish Adaptation, Validity, and Reliability Study of the Fear of Pain Questionnaire (FOPQ-TR)
Brief Title: The Turkish Fear of Pain Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Other Study IDs: 2022-128
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Chronic Headache
Keywords: Chronic headache; Pain related fear; Assessment; Children; validity; cultural adaptation
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Headache Group: Children with chronic headache
- Healthy Group: Children without pain

SUMMARY:
Children's chronic pain is a significant condition that affects roughly 25% of children, with approximately 3% of them requiring intense pain therapy. In the adult literature, various scales have been established to assess fear of pain. When these scales are studied, fear of pain has been shown to have a role in adult chronic pain research, but this topic has gotten less attention in pediatric chronic pain research. The Fear of Pain Questionnaire for Children (FOPQ-C) is a questionnaire that addresses this knowledge gap. The purpose of this study is to determine the validity and clinical utility of the Fear of Pain Questionnaire for Children (FOPQ-C) Scale in the Turkish community.

DETAILED DESCRIPTION:
Pain is a multidimensional experience that includes sensory, cognitive, emotional, and social factors. The International Association for the Study of Pain defines chronic pain as pain that lasts longer than three months, besides the lack of a clear description. Chronic pain is a critical developmental health issue that can be recurring or persistent, causing significant disruption in everyday life. Children with chronic pain that is continuous or recurrent may be unable to attend school, may withdraw from social activities, and may develop internalizing symptoms as a result of their discomfort. Given these findings, researchers and clinicians must focus on concerns connected to pediatric chronic pain in order to reduce these challenges and develop appropriate methods. Adults are reported to suffer from 19 percent of chronic pain, with two-thirds describing their pain as "persistent" and 50% describing it as "unbearable." Chronic pain has emerged as a significant problem in children, affecting around one out of every four children, while approximately 3% of children require intense pain therapy.

Psychosocial factors interact with physiological processes to influence pain outcomes such as pain perception and impairment, according to the biopsychosocial model of chronic pain. Fear of pain is a psychological mechanism that has been shown to be effective in predicting chronic pain and accompanying disability in adults. When pain-related sensations are viewed as dangerous, fear of pain develops. The Fear Avoidance Model of Pain outlines how fear of pain influences the outcomes of people who are in chronic pain. Many elements of the condition, including experimentally generated pain severity, pain during dental treatment, chronic pain behavior, and pain-related disability, have been linked to fear of pain. Simultaneously, in the Fear Avoidance Model of Pain, if pain is seen as threatening, pain-related fear develops, leading to avoidance. Simultaneously, in the Fear Avoidance Model of Pain, if pain is seen as threatening, pain-related fear develops, leading to avoidance behaviors and hypervigilance. After that, there's incapacity and depression. These negative outcomes aggravate the fear and avoidance loop. While assessing fear of pain is critical, assessing fear of re-injury is more difficult because it can entail movement, physical activity, or a mix of these things. Furthermore, patients frequently do not report or subjectively sense pain, but rather have trouble performing the actions or activities that have been required of them.

In the adult literature, various scales have been established to assess fear of pain. Fear of pain has been shown to have a role in adult chronic pain research, but it has gotten less attention in pediatric chronic pain research. The Fear of Pain Questionnaire for children and parents (FOPQ-C SF, FOPQ-P) is a questionnaire that addresses this knowledge gap. As a result, the purpose of this study is to see if the Fear of Pain Questionnaire for Children & Parents (FOPQ-C, FOPQ-P) Scale is valid in the Turkish community and how effective it is in therapeutic practice.

ELIGIBILITY:
Inclusion criteria of children with chronic pain:

(1) Being diagnosed with chronic pain. (2) To have the cognitive ability to answer questions for assessment. (3) Completing the test-retest assessment. (4) To be the native language Turkish.

* Exclusion criteria for children with chronic pain:

  1. Uncontrollable psychological diseases (eg, attention deficit hyperactivity disorder, autism spectrum disorder, schizophrenia, bipolar disorder, major depressive disorder), specific pathologies, will not be included in the study.
  2. Patients who started a new treatment during the study or 6 weeks before the study.
  3. Study participants will be instructed not to take analgesics for 48 hours prior to assessments.

Inclusion criteria for healthy children:

1. between the ages of 5-18.
2. Not having any psychiatric or neurological diagnosis.
3. To be the native language Turkish.

Exclusion criteria for healthy children:

1. Families and children who did not agree to participate in the study.
2. To have received medical treatment for any neuropsychiatric disorder.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with chronic pain at aged 5-18 years and their parents, their health peers without chronic pain and their parents
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-08 (Estimated); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain of fear for children | Baseline
  The Fear of Pain Questionnaire-Short Form (FOPQ-C-SF) for Children is a 10-item variant of the 24-item Fear of Pain Questionnaire for Children. It uses children's self-reports to assess pain-related anxieties (4 items) and avoidance behaviors (6 items). When I'm in pain, for example, I cancel my plans. When I'm in pain, I'm worried something bad may happen. A 0-4 Likert scale is used for scoring. A score of 0 indicates significant disagreement, while a score of 5 indicates great agreement. The total score is calculated by aggregating the individual item scores. Higher pain-related fear and avoidance behavior are associated with higher scores.
Evaluation of pain of fear for parents | Baseline
  The Fear of Pain Scale for Children-Parent Form (FOPQ-P) is a scale that evaluates children's fear of pain with a parent report. FOPQ-P consists of 23 items. The scale assesses fear of pain in three sub-areas. These are: Fear of Pain (8 items), Avoidance of Activities (10 items), and Avoidance of School (5 items). Scoring is done on a Likert scale of 0-4 points. The parent rates the child's approach to pain that has existed for several hours or throughout the day, from 0 = strongly disagree to 4 = strongly agree.

SECONDARY OUTCOMES:
Evaluation of pain catastrophing for children | Baseline
  The Pain Catastrophing Scale was developed to assess adults' pain-related catastrophizing thoughts. The Pain Catastrophizing Scale-Child (PCS-C) is an adapted version of the Pain Catastrophizing Scale for children. PCS-C evaluates catastrophizing behavior with 13 items: thinking long about pain (4 items), magnifying pain (3 items), and helplessness (6 items). For example, I can't get the pain out of my mind. I'm afraid my pain will get worse. There is nothing I can do to reduce the pain. Scoring is done on a Likert scale of 0-4 points. 0=not at all; 4=extremely The adult version of the Turkish version of the Pain Catastrophizing Scale for families will be used.
Evaluation of pain for children | Baseline
  It is a valid and reliable scale that children and their families prefer to use when determining the level of discomfort. It is made up of six different facial expressions that represent the degree of pain. From a happy face (0 points) to a very sad and crying expression, they show the stages of increasing pain (10 points). Each facial expression's meaning is carefully explained to the child. The severity of pain during facials is rated by children.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, Assoc. Prof, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results are going to publish the journal

REFERENCES:
- [Result] Palermo TM, Chambers CT. Parent and family factors in pediatric chronic pain and disability: an integrative approach. Pain. 2005 Dec 15;119(1-3):1-4. doi: 10.1016/j.pain.2005.10.027. Epub 2005 Nov 18. No abstract available. PMID 16298492
- [Result] Palermo TM. Impact of recurrent and chronic pain on child and family daily functioning: a critical review of the literature. J Dev Behav Pediatr. 2000 Feb;21(1):58-69. doi: 10.1097/00004703-200002000-00011. PMID 10706352
- [Result] King S, Chambers CT, Huguet A, MacNevin RC, McGrath PJ, Parker L, MacDonald AJ. The epidemiology of chronic pain in children and adolescents revisited: a systematic review. Pain. 2011 Dec;152(12):2729-2738. doi: 10.1016/j.pain.2011.07.016. PMID 22078064
- [Result] Jiao J, Vincent A, Cha SS, Luedtke CA, Kim CH, Oh TH. Physical Trauma and Infection as Precipitating Factors in Patients with Fibromyalgia. Am J Phys Med Rehabil. 2015 Dec;94(12):1075-82. doi: 10.1097/PHM.0000000000000300. PMID 25888651
- [Result] Hechler T, Dobe M, Zernikow B. Commentary: A worldwide call for multimodal inpatient treatment for children and adolescents suffering from chronic pain and pain-related disability. J Pediatr Psychol. 2010 Mar;35(2):138-40. doi: 10.1093/jpepsy/jsp066. Epub 2009 Aug 14. No abstract available. PMID 19684118
- [Result] Leeuw M, Goossens ME, Linton SJ, Crombez G, Boersma K, Vlaeyen JW. The fear-avoidance model of musculoskeletal pain: current state of scientific evidence. J Behav Med. 2007 Feb;30(1):77-94. doi: 10.1007/s10865-006-9085-0. Epub 2006 Dec 20. PMID 17180640
- [Result] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Result] Berniger Romariz JA, Nonnemacher C, Abreu M, Dickel Segabinazi J, Bandeira JS, Beltran G, Souza A, Torres IL, Caumo W. The Fear of Pain Questionnaire: psychometric properties of a Brazilian version for adolescents and its relationship with brain-derived neurotrophic factor (BDNF). J Pain Res. 2019 Aug 7;12:2487-2502. doi: 10.2147/JPR.S199120. eCollection 2019. PMID 31496790